CLINICAL TRIAL: NCT01416818
Title: A Randomized, Double-Blind, Placebo-Controlled Study of "Xiaoyao Pill" Treatment of Depression in Patients With Parkinson's Disease
Brief Title: Treatment of Depression in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Piu Chan, MD, PhD., Xuanwu Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008XYRCT
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Depression in Parkinson's Disease
Keywords: Depression;; Parkinson's disease;; antidepressant
MeSH Terms: conditions — Depression; Parkinson Disease | interventions — xiaoyao

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- group 1 (Experimental)
  Interventions: Drug: Xiaoyao Pill
- group 2 (Active Comparator)
  Interventions: Drug: Bupleurum+Ginkgo
- group 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Xiaoyao Pill — herb extracts,were received two times a day for 12 weeks without dose changing.
  Arms: group 1
Drug: Bupleurum+Ginkgo — herb extracts, were received two times a day for 12 weeks without dose changing.
  Arms: group 2
Drug: placebo — The placebo looked like herb extracts and were also received two times a day for 12 weeks without dose changing.
  Arms: group 3

SUMMARY:
The goal of this study is to evaluate the efficacy of Traditional Chinese Medicine-"Xiaoyao Pill" (Herb extracts)on depression, compared to placebo and "Bupleurum+Ginkgo" in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Depression as the most common non-motor comorbidity of Parkinson's disease (PD), have a negative impact on disability and quality of life.

Traditional Chinese Medicine has shown effects on several depression. It is not known if TCM also is effective for depression in PD. This study is to investigate "Xiaoyao Pill", an antidepressant in TCM, on depression in PD.

A total of 60 patients with depression in PD will be randomized to each of the three arms.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease without dementia
* Depression
* Males or females
* Willing and able to give informed consent

Exclusion Criteria:

* cognitive dysfunction
* other serious diseases

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale | 12 weeks
  Change of Hamilton Depression Scale score on week 12 from baseline.

SECONDARY OUTCOMES:
the responder rate (defined as score reduction of HAMD-17>=50%) | 12 weeks
the Geriatric Depression Scale | 12 weeks
  GDS-30

CONTACTS AND LOCATIONS:
Overall Officials: Piu Chan, MD. PhD., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, China